CLINICAL TRIAL: NCT03699384
Title: A Phase I/II Safety and Clinical Activity Study of Combination Azacitidine and Avelumab in Patients With Acute Myeloid Leukemia (AML) and Minimal Residual Disease (MRD)
Brief Title: Safety and Clinical Activity Study of Combination Azacitidine and Avelumab in Patients With Acute Myeloid Leukemia (AML) and Minimal Residual Disease (MRD)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study sponsor discontinued support
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-012
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Acute Myeloid Leukemia (AML); Minimal Residual Disease
Keywords: Azacitidine; Avelumab; 18-012
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Azacitidine; avelumab

STUDY DESIGN:
Intervention Model Description: This is an open label, phase I/II prospective clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine and Avelumab (Experimental): All enrolled patients will receive 1 cycle of AZA followed by cycles of combination AZA+Avelumab.
  Interventions: Drug: Azacitidine; Drug: Avelumab

INTERVENTIONS:
Drug: Azacitidine — AZA 75 mg/m^2 SC or IV D 1-7 28 day cycle x 1
Drug: Avelumab — Avelumab 10mg/kg IV D1, D15, 28d cycle Until progression or MRD If MRD-, tx x 1 yr or go to allo SCT

SUMMARY:
This is a phase I / II study. The purposes of this study are to: 1) find out what effects, good and/or bad, the combination of the experimental drug avelumab and the drug azacitidine has on people with AML and MRD, and 2) test if the two drugs, avelumab and azacitidine, are effective in getting rid of AML MRD when the drugs are given together in combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 years of age.
* Subjects must have a history of AML as defined by WHO criteria. AML patients with any cytogenetic abnormalities are eligible except for patients with t (15;17) (acute promyelocytic leukemia). AML patients who have never undergone allogeneic stem cell transplant must have adverse-risk AML by ELN criteria77 to be eligible. Patients with a history of therapy related AML, myeloid sarcoma, or patients whose AML evolved from an antecedent MDS or MPN are also eligible. Patients with any molecular mutations are eligible.
* Subjects must have received therapy for AML and have a bone marrow biopsy within 28 days prior to registration that demonstrates a morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) as defined by European Leukemia Net (ELN) criteria. Patients with prior myeloid sarcoma must have no residual evidence of extramedullary leukemia.
* Subjects may have received any prior therapy for AML including cytotoxic agents, hypomethylating agents, or other therapeutics to achieve morphologic CR or CRi.
* Subjects must have MRD in a bone marrow aspirate within 28 days prior to registration from the same bone marrow sample which demonstrates morphologic CR. MRD is identified by multiparameter flow cytometry as a cell population showing deviation from normal antigen-expression patterns seen in specific cell lineages at specific stages of maturation. Any level of residual flow cytometric disease is considered MRD positive.
* Subjects must be amenable to serial bone marrow biopsies, peripheral blood sampling, and urine sampling during the study.
* Subjects or their legal representatives must be able to understand and sign an informed consent.
* Subjects must have ECOG PS of 0 to 2. 9. Subjects must have adequate hematological function defined by absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L, platelet count ≥ 50 × 10^9/L, and hemoglobin ≥ 9 g/dL (may have been transfused)
* Subjects must have adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN
* Subjects must have adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula
* Subjects must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer. (Subjects with residual Grade 1-2 toxicity, for example Grade 1-2 peripheral neuropathy or residual alopecia, are allowed with approval of the principal investigator.)
* Negative serum pregnancy test at screening for women of childbearing potential.
* Subjects must use highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1% per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after avelumab treatment.)

Exclusion Criteria:

* Patients with prior allogeneic stem cell transplantation (SCT) who have had:

  1. allo-SCT performed <3 months prior to enrollment; or
  2. immunosuppressive treatment for acute or chronic graft-versus-host disease (GVHD) within 3 months prior to enrollment (with the exception of those patients who required ≤15 mg/day oral prednisone or equivalent); or
  3. acute Grade 3 or Grade 4 GVHD at any time in the past (as defined by the modified Seattle Glucksberg Criteria); or
  4. prior chronic GVHD (as defined by the NIH Consensus Development Project), persisting for >6 months, which required systemic immunosuppression (with the exception of those patients who required ≤15 mg/day oral prednisone or equivalent); or
  5. a donor lymphocyte infusion (DLI) within 6 months prior to enrollment; or
  6. is currently on treatment with GVHD prophylaxis medications tacrolimus, sirolimus, or cyclosporine
* Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
* Significant acute or chronic infections including, among others:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

  1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
  2. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
  3. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable
  4. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) are acceptable.
* Known severe hypersensitivity reactions to Azacitidine or to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia, vitiligo, and sensory neuropathy Grade ≤ 2 is acceptable

  a. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with Avelumab and/or Azacitidine (e.g., hearing loss) may be included after consultation with the Study Physician.
* Pregnancy or lactation
* Known alcohol or drug abuse
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject"s tolerance of trial treatment
* Subjects with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject"s ability to sign informed consent, cooperate, or participate in the study.
* Vaccination within 4 weeks of the first dose of Azacitidine and while on trial is prohibited except for administration of inactivated vaccines
* History of idiopathic pulmonary fibrosis, organizing pneumonitis (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis
* Subjects who have previously received immune checkpoint blockade are excluded unless they meet the following conditions:

  1. Last dose of immunotherapy must have been administered at least 100 days prior to planned first dose of Azacitidine;
  2. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy;
  3. All AEs while receiving prior immunotherapy must have resolved to ≤ Grade 1 or baseline prior to screening for this study. Must not have experienced a ≥ Grade 3 AE or neurologic or ocular AE of any grade; Note: Subjects with endocrine AE of any grade are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic;
  4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
* Subjects who received systemic anticancer therapy or radiotherapy <14 days prior to their first day of Azacitidine.
* Subjects who received a small molecule investigational agent <14 days prior to their first day of Azacitidine.
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of investigational product(s).
* Subjects with an active severe infection or with an unexplained fever >38.5°C during screening visits or on their first day of study drug administration.
* Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of C1D1.
* Subjects with a history of myocardial infarction within the last 6 months.
* Subjects with uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg or diastolic BP >100 mmHg) are excluded. Subjects requiring 2 or more medications to control hypertension are eligible with principal investigator approval.
* Subjects with known unstable or uncontrolled angina pectoris.
* Subjects with ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥ 2 or prolongation of the QTc interval to >500 msec.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product(s) or interpretation of subject safety or study results.
* Subjects with favorable risk or intermediate-risk AML by ELN criteria (see appendix B) who have MRD but who have never undergone allogeneic SCT are excluded. Patients with AML who have MRD after allogeneic SCT are allowed regardless of initial AML risk status provided they are otherwise eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities as assessed by CTCAE v4.0 | 1 year
  Up to 6 pre-allo SCT patients who are evaluable for DLT will be enrolled, with the first 3 patients enrolled in a sequential manner with a 1-week interval between the start of dosing for each patient. If the regimen appears tolerable in the first 3 patients (i.e., ≤ 1 of the first 3 patients enrolled experiences a DLT), then the next 3 patients will be enrolled concurrently. If more than 1 out of 6 in the pre-alloSCT group has a DLT, the trial will stop accrual. The combination will be considered safe in pre-allo SCT patients if one or no patient has a DLT out of the six patients. If the combination is safe in pre-alloSCT patients, additional pre-alloSCT patients will begin enrollment for the expanded phase II portion of the study, and accrual of 6 post-alloSCT patients for separate safety evaluation will begin. Toxicity will be graded on a scale of 1 to 5 as described by the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
sustained MRD negativity (Phase II) | 1 year
  This is defined as the time from the first dose of azacitidine to a patient"s confirmed MRD negativity on the second bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Goldberg, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm